CLINICAL TRIAL: NCT04639947
Title: Reliability and Reproducibility of the Eye Check Tonometer Pressure Measurements as Measured by Patients Reliability and Reproducibility of the Eye Check Tonometer Pressure Measurements as Measured by Patients
Brief Title: Reliability and Reproducibility of the Eye Check Tonometer
Acronym: EyeCheck
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to low accrual
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00106897
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Glaucoma; Glaucoma, Suspect
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Intervention Model Description: All subjects will first take their pressure using the EyeCheck with contact lens in and then remove their lens have pressures taken with Goldmann and Tonopen (two standard of care techniques of taking pressures of the eyes).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- EyeCheck (Experimental): EyeCheck pressures will be measured with contact lens in place
  Interventions: Device: EyeCheck
- Traditional Tonometer (Goldmann and Tonopen) (Active Comparator): Pressures will be measured with both Goldmann and Tonopen (both traditional tonometers to take the intraocular pressure (IOP) measurements of the eye).
  Interventions: Device: Traditional Tonometer (Goldmann and Tonopen)

INTERVENTIONS:
Device: EyeCheck — EyeCheck is a newly developed device to provide intraocular pressure (IOP) measurements of the eyes.
  Arms: EyeCheck
Device: Traditional Tonometer (Goldmann and Tonopen) — Standard of care intraocular pressures will be taken using the Goldmann and Tonopen to compare to the EyeCheck.
  Arms: Traditional Tonometer (Goldmann and Tonopen)

SUMMARY:
To investigate whether the new applanation tonometer (EyeCheck monitor) can provide intraocular pressure (IOP) measurements comparable to those of traditional tonometers such as the Goldmann applanation tonometer and the Tonopen.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older,
* Any glaucoma patient or glaucoma suspect patient
* Presents for an appointment wearing their own soft contact lens.

Exclusion Criteria:

* Arthritis affecting the upper extremity in the patient or caregiver
* Patient unwilling or assessed to be unable to comply with the study protocol
* Any corneal abnormalities such as opacities, scars, Fuchs dystrophy, map dot fingerprint dystrophy, history of recurrent corneal abrasion, corneal surgery such as Lasik, PRK, DSAEK, transplant or implant
* History of any ongoing ocular symptoms such as eye pain or redness or discharge
* History of recent ocular surgery (done in the past 3 months)
* History of a any filtering or tube surgery for glaucoma (to reduce risk of infection associated complications)
* Recent eye infection (within the past 3 months)
* History of diabetes for > 5 years duration
* Monocular patient
* Best corrected visual acuity< 20/70
* Head or hand tremors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Asrani, MD, Principal Investigator — Duke Eye Center
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Currently, there is no plan to share data with other researchers.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each study participant was enrolled into both arms. Therefore 22 subjects were enrolled and had testing in each arm.
Units Other Than Participants: eyes
Groups:
- EyeCheck and Traditional Tonometer (Goldmann and Tonopen): EyeCheck pressures will be measured with contact lens in place
  EyeCheck: EyeCheck is a newly developed device to provide intraocular pressure (IOP) measurements of the eyes.
  Pressures will be measured with both Goldmann and Tonopen (both traditional tonometers to take the intraocular pressure (IOP) measurements of the eye).
  Traditional Tonometer (Goldmann and Tonopen): Standard of care intraocular pressures will be taken using the Goldmann and Tonopen to compare to the EyeCheck.
Period: Overall Study
Arm/Group | EyeCheck and Traditional Tonometer (Goldmann and Tonopen)
Started | 22; 22 eyes
Completed | 21; 21 eyes
Not Completed | 1; 1 eyes
Not completed — Screen fail | 1

BASELINE CHARACTERISTICS:
Arm/Group | EyeCheck and Traditional Tonometer (Goldmann and Tonopen)
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 14
Age, Continuous [Mean (Full Range); unit: years] | 67 [37 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP) Measurements
Description: Compare EyeCheck intraocular pressure (IOP) measurements comparable to those of traditional tonometers (Goldmann and tonopen)
Time Frame: Baseline
Population: Participants received both EyeCheck and traditional tonometer measurements.
Measure: Mean (Full Range); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | EyeCheck | Traditional Tonometer (Goldmann and Tonopen)
Number analyzed (Participants) | 22 | 22
Number analyzed (eyes) | 22 | 22
mmHg | 17.4 [10 to 26] | 19.1 [13 to 25]

ADVERSE EVENTS:
Time Frame: 1 day
Description: Each study participant was enrolled into both arms.
Arm/Group | EyeCheck | Traditional Tonometer (Goldmann and Tonopen)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT04639947/Prot_SAP_001.pdf